CLINICAL TRIAL: NCT03536949
Title: A Randomized, Double-Masked, Placebo-Controlled Phase 3 Study of the Safety of RVL-1201 in the Treatment of Acquired Blepharoptosis (Study RVL-1201-203)
Brief Title: Study of Safety of RVL-1201 in Treatment of Blepharoptosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RVL-1201-203
Record Dates: First submitted 2018-04-11; First posted 2018-05-25 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RVL-1201 Ophthalmic Solution, 0.1% (Experimental): RVL-1201 (oxymetazoline hydrochloride) ophthalmic solution 0.1%
  Interventions: Drug: RVL-1201
- Vehicle ophthalmic solution (Placebo Comparator): Vehicle placebo ophthalmic solution
  Interventions: Other: Vehicle ophthalmic solution

INTERVENTIONS:
Drug: RVL-1201 — RVL-1201 ophthalmic solution, 0.1%
  Arms: RVL-1201 Ophthalmic Solution, 0.1%
Other: Vehicle ophthalmic solution — Vehicle placebo ophthalmic solution
  Arms: Vehicle ophthalmic solution

SUMMARY:
Phase 3 study to evaluate the extended safety of RVL-1201 compared to placebo for treatment of blepharoptosis. Eligible subjects will be randomized to one of 2 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 9 years of age or older
2. Females must not be pregnant or planning to get pregnant and must use acceptable form of contraception
3. Must be able to self-administer study medication
4. Must be able to understand and sign an Informed Consent Form (ICF). For minor subjects, the subject's parent or legal guardian must provide permission by signing an ICF on behalf of the subject and the subject should provide assent.

Exclusion Criteria:

1. Congenital ptosis
2. Horner syndrome
3. Myasthenia gravis
4. Mechanical ptosis
5. Previous ptosis surgery
6. Resting heart rate outside the normal range
7. Hypertension with resting diastolic blood pressure
8. Pregnancy or lactation

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Barnet, Dulany Perkins, Phoenix, Arizona
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - North Valley Eye Medical, Mission Hills, California
  - Eye Research Foundation, Newport Beach, California
  - Pendelton Eye Center, Oceanside, California
  - North Bay Eye Associates, Petaluma, California
  - Michael K. Tran, MD Inc., Westminster, California
  - Danbury Eye Physicians and Surgeons, Danbury, Connecticut
  - Hernando Eye Institute, Brooksville, Florida
  - Shettle Eye Research, Largo, Florida
  - West Coast Eye Institute, Lecanto, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center, Maitland, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Coastal Research Associates, Roswell, Georgia
  - Kennar Eye Care, Pittsburg, Kansas
  - Heart of America Eye Care, Shawnee Mission, Kansas
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Mississippi Eye Associates, Ocean Springs, Mississippi
  - Silverstein Eye Centers, Kansas City, Missouri
  - Comprehensive Eye Care, Washington, Missouri
  - Rochester Ophthalmological Group, Rochester, New York
  - South Shore Eye Care, Wantagh, New York
  - CEENTA, Charlotte, North Carolina
  - Cornerstone Eye Care, High Point, North Carolina
  - Drs. Quinn, Foster & Associates, Athens, Ohio
  - Apex Eye, Cincinnati, Ohio
  - Abrams Eye Center, Cleveland, Ohio
  - Nashville Vision Associates, Nashville, Tennessee
  - Round Rock Eye Consultants, Austin, Texas
  - Texan Eye / Keystone Research, Ltd., Austin, Texas
  - Lake Travis Eye and Laser Center, Lakeway, Texas
  - R & R Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned sample size approximately 225 subjects, 150 subjects in the RVL-1201 group and 75 subjects in the Vehicle group, to be enrolled at approximately 30 clinical sites in the U.S.
Groups:
- RVL-1201 Ophthalmic Solution, 0.1%: RVL-1201 (oxymetazoline hydrochloride) ophthalmic solution 0.1% One drop each eye QD for 84 days
- Vehicle Ophthalmic Solution: Vehicle placebo ophthalmic solution One drop each eye QD for 84 days
Period: Overall Study
Arm/Group | RVL-1201 Ophthalmic Solution, 0.1% | Vehicle Ophthalmic Solution
Started | 157 | 77
Completed | 143 | 75
Not Completed | 14 | 2
Not completed — Adverse Event | 4 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Non-compliance | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | RVL-1201 Ophthalmic Solution, 0.1% | Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 157 | 77 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 65 | 38 | 103
  >=65 years | 90 | 38 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (14.64) | 63.3 (14.63) | 63.6 (14.60)
Age, Customized [Median (Full Range); unit: years] | 66 [13 to 90] | 64 [15 to 90] | 66 [13 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 53 | 179
  Male | 31 | 24 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 5 | 19
  Not Hispanic or Latino | 143 | 72 | 215
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 12 | 8 | 20
  White | 137 | 66 | 203
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 157 | 77 | 234

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Intraocular Pressure (IOP) at Day 84
Description: Intraocular pressure will be measured in mmHg utilizing a tonometer and using the standard of care. If possible, the same calibrated instrument should be used for a given subject throughout the study.
Time Frame: Screening/Day 1 to Day 84
Population: The safety population includes all subjects who receive at least one dose of double-masked study treatment and have at least one post-dose visit.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- RVL-1201 Ophthalmic Solution, 0.1%: Participants with Acquired Blepharoptosis administered 1 drop of RVL-1201 in each eye once daily
- Vehicle Ophthalmic Solution: Participants with Acquired Blepharoptosis administered 1 drop of Vehicle in each eye once daily
Arm/Group | RVL-1201 Ophthalmic Solution, 0.1% | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 157 | 77
mmHg
  Mean Change from Baseline IOP (OD) | -0.6 (2.40) | -0.2 (2.52)
  Mean Change from Baseline IOP (OS) | -0.6 (2.42) | -0.2 (0.41)

2. Primary Outcome: Mean Change From Baseline in Pupil Diameter (PD) at Day 84
Description: Pupil diameter will be measured in millimeters (either horizontally or vertically if top of pupil is not visible in photograph) from the external photograph.
Time Frame: Screening/Day 1 to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | RVL-1201 Ophthalmic Solution, 0.1% | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 157 | 77
Millimeters (mm)
  Mean Change From Baseline PD (OD) | 0.0 (0.77) | -0.1 (0.66)
  Mean Change from Baseline PD (OS) | 0.0 (0.77) | -0.1 (0.59)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were assessed at Baseline through Day 84 (end of study).
Description: AEs spontaneously reported by the subject and/or in response to an open questions from the study personnel or revealed by observation were recorded in the electronic Case Report Form (eCRF).
Arm/Group | RVL-1201 Ophthalmic Solution, 0.1% | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/77
Serious Adverse Events (participants affected / at risk) | 2/157 | 0/77
Other Adverse Events (participants affected / at risk) | 19/157 | 5/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVL-1201 Ophthalmic Solution, 0.1% (N=157) | Vehicle Ophthalmic Solution (N=77)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVL-1201 Ophthalmic Solution, 0.1% (N=157) | Vehicle Ophthalmic Solution (N=77)
Dry eye (Eye disorders) | 7 (12) | 1 (2)
Conjunctival hyperaemia (Eye disorders) | 5 (9) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Vital dye staining cornea present (Investigations) | 5 (7) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT03536949/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03536949/SAP_001.pdf